CLINICAL TRIAL: NCT06457165
Title: Predicting Difficult Intubation in Obese Patients: The Role of Anthropometric Measurements and Ultrasonograpic Suprasternal Adipose Tissue Thickness
Brief Title: The Role of Anthropometric Measurements and Ultrasonograpic Suprasternal Adipose Tissue Thickness
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayça Özcan, Assoc. Prof. MD, Ankara City Hospital Bilkent
Other Study IDs: Difficult Intubation
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Intubation; Difficult or Failed; Obesity; Anesthesia
MeSH Terms: conditions — Obesity | interventions — Waist Circumference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult Intubation: Abdominal circumference, waist circumference, arm circumference, distance between incisions,TMD and SMD measurements, Mallampati test, Wilson score, and suprasternal subcutaneous adipose tissue thickness were measured and recorded. ECG, SBP and DBP, and SpO2 monitoring were performed. Pre-oxygenation was performed using a 100% oxygen face mask for 3 min before the induction of anesthesia. Induction of anesthesia was achieved with IV 1 mg/kg lidocaine, 0.125 mcgr/kg fentanyl, 2 mg/kg propofol, and 0.6 mg/kg rocuronium bromide. After 2 min of adequate muscle relaxation, the patient was intubated with an endotracheal tube of appropriate diameter. Cormack-Lehane score was evaluated during laryngoscopy. Patients with more than 3 intubation attempts by an experienced anesthesiologist were considered difficult to intubate. In maintenance, 0.1 mcg/kg/h remifentanil was administered in sevoflurane O2-air mixture.
  Age, sex, body weight,BMI, and ASA scores were recorded.
  Interventions: Device: Difficult Intubation; Device: Not Difficult Intubation
- Not Difficult Intubation: Abdominal circumference, waist circumference, arm circumference, distance between incisions,TMD and SMD measurements, Mallampati test, Wilson score, and suprasternal subcutaneous adipose tissue thickness were measured and recorded. ECG, SBP and DBP, and SpO2 monitoring were performed. Pre-oxygenation was performed using a 100% oxygen face mask for 3 min before the induction of anesthesia. Induction of anesthesia was achieved with IV 1 mg/kg lidocaine, 0.125 mcgr/kg fentanyl, 2 mg/kg propofol, and 0.6 mg/kg rocuronium bromide. After 2 min of adequate muscle relaxation, the patient was intubated with an endotracheal tube of appropriate diameter. Cormack-Lehane score was evaluated during laryngoscopy. Patients with more than 3 intubation attempts by an experienced anesthesiologist were considered difficult to intubate. In maintenance, 0.1 mcg/kg/h remifentanil was administered in sevoflurane O2-air mixture.
  Age, sex, body weight,BMI, and ASA scores were recorded.
  Interventions: Device: Difficult Intubation; Device: Not Difficult Intubation

INTERVENTIONS:
Device: Difficult Intubation — Noted for each patient.
  Other Names: Age; ASA; BMI; Arm circumference; TMD; SMD; Distance between incisions; Abdominal circumference; Waist circumference; Suprasternal adipose tissue thickness; Mallampati; Cormack-Lehane score; Wilson score
Device: Not Difficult Intubation — Noted for each patient.
  Other Names: Age; ASA; BMI; Arm circumference; TMD; SMD; Distance between incisions; Abdominal circumference; Waist circumference; Suprasternal adipose tissue thickness; Mallampati; Cormack-Lehane score; Wilson score

SUMMARY:
Prediction of difficult preoperative intubation in obese patients and completion of preparations for difficult intubation both reduce the risk of repeated intubation and prevent complications.

In this study, the investigators aimed to evaluate whether anthropometric measurements are superior in defining difficult preoperative airways.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines obesity, the incidence of which has increased significantly worldwide and is one of the important causes of difficult airway in terms of anesthesia, as obesity when the body mass index (BMI) is above 30. Access to the upper airway is difficult in obese patients, in whom excessive adipose tissue accumulates in the breast, neck, chest, and abdomen. Determining preoperative difficult intubation parameters in obese patients and entering the case preparation both reduce the risk of repeated intubation and prevent intraoperative and postoperative complications.

However, there are still insufficient tests to predict difficult intubation. Many studies have shown that multiple factors such as Mallampati score, high body mass index (BMI), increased neck circumference, and the ratio of neck circumference to thyromental distance are predictors of difficult intubation in obese patients. The introduction of ultrasonography into daily use has led to the use of ultrasonographic parameters in predicting difficult intubation and laryngoscopy. In this study, the investigators aimed to evaluate whether ultrasonography is useful in defining difficult preoperative airways, in addition to anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* ASA 1-3
* BMI ≥30 kg/m2
* ASA 1-3
* Scheduled for elective abdominal surgery under general anesthesia

Exclusion Criteria:

* <18 and >60 years
* ASA>3
* BMI<30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 40 patients between the ages of 18-60 years, ASA 1-3, BMI ≥30 kg/m2, ASA 1-3, scheduled for elective abdominal surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Suprasternal Adipose Tissue Thickness | within 10 minutes before going into surgery
  It is predicted that it may indicate difficult intubation.

SECONDARY OUTCOMES:
Abdominal circumference | within 10 minutes before going into surgery
  Noted for each patient.
Waist circumference | within 10 minutes before going into surgery
  Noted for each patient.
Arm circumference | within 10 minutes before going into surgery
  Noted for each patient.
Distance between incisions | within 10 minutes before going into surgery
  Noted for each patient.
Thyromental distance measurement | within 10 minutes before going into surgery
  Noted for each patient.
Sternomental distance measurement | within 10 minutes before going into surgery
  Noted for each patient.
Mallampati Score | within 10 minutes before going into surgery(class 1-4; 1 means good and 4 means bad)
  Noted for each patient.
Wilson score | within 10 minutes before going into surgery(grade 0-10; 0 means good, 10 means bad)
  Noted for each patient.
Cormack-Lehane score | 1. minute after intubation(class 1-4; 1 means good and 4 means bad)
  Noted for each patient.
Age | within 10 minutes before going into surgery
  Noted for each patient.
Sex | within 10 minutes before going into surgery
  Noted for each patient.
ASA | within 10 minutes before going into surgery(grades 1-6; 1 means good and 6 means bad)
  Noted for each patient.
BMI | within 10 minutes before going into surgery
  Noted for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Tuba Dumanlı Özcan, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)